CLINICAL TRIAL: NCT07084532
Title: The Effect of Chewing Gum on Dry Mouth in Individuals With Diabetes Mellitus
Brief Title: Effects of Chewing Gum for Dry Mouth in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Saadet Aybek,, Clinical Nurse, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CankırıKU-SBF-SA-01
Record Dates: First submitted 2025-06-13; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Diabetes (DM); Dry Mouth
Keywords: Diabetes Mellitus; Dry Mouth; Chewing Gum; Nursing Care
MeSH Terms: conditions — Diabetes Mellitus; Xerostomia | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: Quasi-experimental in a pre-test-post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group was informed about the study. Dry mouth was noted at baseline. Individuals in the intervention group were asked to chew sugarless gum for 15 minutes before meals and before 3 main meals for 7 days.
  Interventions: Other: Chewing gum
- Standart Therapy Group (Experimental): Patients in the control group were also informed about the study and completed a data collection form via face-to-face interview. No interventions were performed on the control group patients. They were also informed that they would be re-evaluated one week later during the study and were asked to refrain from chewing gum during this period.
  Interventions: Other: Standart therapy group

INTERVENTIONS:
Other: Chewing gum — Dry mouth was diagnosed in the initial assessment of diabetic individuals assigned to the intervention group. Following the assessment, they were asked to chew gum for 15 minutes before each main meal for seven days. Dry mouth was re-evaluated with the Xerostomia Scale seven days later.
  Arms: Intervention Group
Other: Standart therapy group — The control group was informed about the study. They were then assessed for dry mouth. They were asked to follow their standard treatment. They were warned not to chew gum. A day later, dry mouth was assessed again without any treatment.
  Arms: Standart Therapy Group

SUMMARY:
Dry mouth can seriously affect the quality of life of individuals because it affects chewing and swallowing functions. One of the diseases in which dry mouth occurs as a side effect of many diseases and/or treatments is diabetes mellitus. The aim of this study was to determine the effect of chewing gum on dry mouth in individuals with diabetes mellitus.

DETAILED DESCRIPTION:
Diabetic autonomic neuropathy and microvascular changes in the oral mucosa are thought to cause decreased salivary secretion in individuals. Furthermore, poor blood glucose regulation and the accompanying polyuria can cause dehydration, leading to dry mouth and decreased salivary secretion. Decreased salivary secretion and subsequent changes in the oral mucosa have been reported in diabetic individuals with poor glycemic control.

Chewing gum is one of the activities that increases salivary secretion. It affects salivary pH and flow rate through both taste and mechanical stimulation, relieving dry mouth symptoms in individuals. While the unstimulated salivary flow rate in humans is 0.3 ml/min, this rate can reach 7 ml/min in someone chewing gum. Due to these known properties, chewing gum can be beneficial for dry mouth in individuals.

Literature reviews have shown that chewing gum reduces the feeling of dry mouth, increases salivary secretion, and quenches thirst. It is also believed that increased salivary secretion dilutes the bacterial load in the mouth, thus reducing the risk of periodontal disease. It is anticipated that chewing gum may be a factor that can improve the quality of life for patients with chronic diseases that require fluid restriction and a special diet. A review of the literature found no studies demonstrating the effect of gum chewing on dry mouth in individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for individuals in the study were; being diagnosed with type 2 diabetes mellitus, having an HbA1c value of 7% and above, being able to communicate verbally, not having hearing loss, and accepting the voluntary consent form voluntarily.

Exclusion Criteria:

* The exclusion criteria for individuals to be included in the study were having additional diseases that caused dry mouth and oral problems and/or using medication or other treatments for this reason (chemotherapy, radiotherapy, Sjögren syndrome, patients who cannot communicate verbally, have hearing problems, do not want to chew gum, use of antihypertensive, anxiolytic and diuretic drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Improvement in dry mouth in individuals with diabetes | 5
  The level of dry mouth of the individuals before and after the intervention was defined by the Xerostomia scale. The scale consists of 11 questions. The lowest possible score is 11 and the highest is 55, with higher scores indicating increased dry mouth.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27478847/